CLINICAL TRIAL: NCT04344847
Title: Incidental Finding of Gastrointestinal Stromal Tumors (GISTs) During Laparoscopic Sleeve Gastrectomy, How to Deal? How Much Safety Margin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bassem Mohamed Sieda (Other Government)
Responsible Party: Sponsor-Investigator, Bassem Mohamed Sieda, Assistant professor of general surgery, faculty of medicine, Zagazig University
Organization: Zagazig University (Other Government)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0000-0002-9590
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Excision Margin
Keywords: Gastrointestinal stromal tumour; Coincidental GIST with LSG; Gastric GIST
MeSH Terms: conditions — Margins of Excision; Gastrointestinal Stromal Tumors

STUDY DESIGN:
Intervention Model Description: With institutional review board approval from Zagazig University Hospitals 338. A double-centre prospective study was conducted on prospectively collected data of all morbidly. 17 patients in Zagazig University Hospitals, Faculty of Medicine, Egypt and 321 patients done in bariatric surgery excellence unit in a tertiary hospital in Riyadh-KSA.
Masking Description: With institutional review board approval from Zagazig University Hospitals 338. A double-centre prospective study was conducted on prospectively collected data of all morbidly. 17 patients in Zagazig University Hospitals, Faculty of Medicine, Egypt and 321 patients done in bariatric surgery excellence unit in a tertiary hospital in Riyadh-KSA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- coincidental GIST during LSG patients (Other): With institutional review board approval from Zagazig University Hospitals 338. A double-centre prospective study was conducted on prospectively collected data of all morbidly. 17 patients in Zagazig University Hospitals, Faculty of Medicine, Egypt and 321 patients done in bariatric surgery excellence unit in a tertiary hospital in Riyadh-KSA.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Excision of Gastric GIST along fundus or body of stomach in the same specimen of LSG with safety margin 1-2cm

SUMMARY:
LSG is thought to be the best choice for obese patients with conincidental GISTs, as a tumour can be resected along with resecting the stomach within the same procedure. The primary endpoint is that, how much does GIST suppose to be far from a staple line to do safe laparoscopic sleeve gastrectomy

DETAILED DESCRIPTION:
The incidence of unsuspected GIST in LSG specimens in our series was high in comparison to cases reported in the literature.

GISTs could be safely removed laparoscopically during LSG surgery with negative microscopic resection margins, with 1-2cm safety margin. Margins less than 1cm, high mitotic rate are adverse prognostic factors.

Examining the whole stomach before resection is mandatory and can easily be done during LSG, GIST can be removed safely with LSG

ELIGIBILITY:
Inclusion Criteria:

All morbid obese patients with BMI more than 35

Exclusion Criteria:

* previous gastric surgery
* patients with hiatus hernia
* age under 21 years

Ages: 21 Years to 42 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 338 (Estimated)
Dates: Start 2016-12-12 (Actual); Primary Completion 2020-05-13 (Estimated); Study Completion 2020-06-12 (Estimated)

PRIMARY OUTCOMES:
Excision of GIST during LSG | 4 years from start of study
  we analyzed the incidence of GISTs in patients underwent LSG and investigated whether simultaneous resection can be oncologically adequate. as long as GIST is distal to staple line with a negative margin, laparoscopic sleeve gastrectomy can be done safely.

CONTACTS AND LOCATIONS:
Locations (1):
- Saudi german hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
WHEN REGISTERED AND APPROVED FOR PUBLICATION, I WILL SHARE THROUGH ALL SCIENTIFIC SITES
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 4 YEARS ,STARTING DECEMBER 2016
Access Criteria: GIST during LSG

REFERENCES:
- [Result] Lyros O, Moulla Y, Mehdorn M, Schierle K, Sucher R, Dietrich A. Coincidental Detection of Gastrointestinal Stromal Tumors During Laparoscopic Bariatric Procedures-Data and Treatment Strategy of a German Reference Center. Obes Surg. 2019 Jun;29(6):1858-1866. doi: 10.1007/s11695-019-03782-y. PMID 30875013
- [Result] Mazer L, Worth P, Visser B. Minimally invasive options for gastrointestinal stromal tumors of the stomach. Surg Endosc. 2021 Mar;35(3):1324-1330. doi: 10.1007/s00464-020-07510-x. Epub 2020 Mar 27. PMID 32221752
- [Result] Inaba CS, Dosch A, Koh CY, Sujatha-Bhaskar S, Pejcinovska M, Smith BR, Nguyen NT. Laparoscopic versus open resection of gastrointestinal stromal tumors: survival outcomes from the NCDB. Surg Endosc. 2019 Mar;33(3):923-932. doi: 10.1007/s00464-018-6393-8. Epub 2018 Aug 31. PMID 30171396